CLINICAL TRIAL: NCT06999980
Title: A Phase II, Multicentre, Parallel Group, Open Label, Randomised Clinical Trial of Neoadjuvant Nivolumab and Ipilimumab Combined With Relatlimab for Patients With Resectable Advanced Melanoma Identified as Poor Responders to Immunotherapy
Brief Title: Neo IRENIE (NEOadjuvant Ipilimumab, RElatlimab, NIvolumab Evaluation)
Acronym: Neo IRENIE
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Melanoma Institute Australia (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MIA2025/522; CA224-1100 (Other: Bristol Myers Squibb)
Record Dates: First submitted 2025-05-23; First posted 2025-05-31 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Cutaneous Melanoma; Mucosal Melanoma
Keywords: Neoadjuvant; Immunotherapy; Randomised trial; Low Responder
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab; Nivolumab; relatlimab; pembrolizumab

STUDY DESIGN:
Intervention Model Description: Phase 2, multicentre, 3 parallel cohorts, open label, randomised clinical trial of neoadjuvant therapy and using a multi-omic predictive biomarker test to identify patients with a 'high' or 'poor' likelihood of response to immunotherapy in one of the cohorts.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Treatment Arm A (Experimental): Ipilimumab at 3 mg per kg with nivolumab at 1 mg per kg will be administered on days 1 and 22 (Q3W) in the neoadjuvant period for a total of 2 doses.
  Interventions: Drug: Ipilimumab 3mg/kg and nivolumab 1mg/kg
- Treatment Arm B (Experimental): Ipilimumab 1mg per kg and the fixed dose combination nivolumab 480 mg and relatlimab 160 mg will be administered on days 1 and 29 (Q4W) for a total of 2 doses.
  Interventions: Drug: Ipilimumab 1mg/kg Nivolumab 480mg and relatlimab 160mg
- Treatment Arm C (Experimental): Fixed dose combination of nivolumab 480 mg and relatlimab 160 mg alone, to be administered on days 1 and 29 (Q4W) for a total of 2 doses.
  Interventions: Drug: Nivolumab 480mg and relatlimab 160mg
- Treatment Arm D (Cohort 1a) (Active Comparator): Ipilimumab at 1 mg per kg with nivolumab at 3 mg per kg will be administered on days 1 and 22 (Q3W) in the neoadjuvant period for a total of 2 doses.
  Interventions: Drug: Ipilimumab 1mg/kg and nivolumab 3mg/kg
- Treatment Arm E (Cohort 1b) (Active Comparator): Ipilimumab at 1 mg per kg with nivolumab at 3 mg per kg will be administered on days 1 and 22 (Q3W) in the neoadjuvant period for a total of 2 doses.
  Interventions: Drug: Ipilimumab 1mg/kg and nivolumab 3mg/kg
- Treatment Arm F (Active Comparator): Pembrolizumab 200 mg will be administered on days 1 and 22 (Q3W) in the neoadjuvant period for a total of 2 doses
  Interventions: Drug: Pembrolizumab 200 mg

INTERVENTIONS:
Drug: Ipilimumab 3mg/kg and nivolumab 1mg/kg — Neoadjuvant for 2 doses on days 1 and 22
  Other Names: Arm A
  Arms: Treatment Arm A
Drug: Ipilimumab 1mg/kg Nivolumab 480mg and relatlimab 160mg — Neoadjuvant for 2 doses at days 1 and 29
  Other Names: Arm B
  Arms: Treatment Arm B
Drug: Nivolumab 480mg and relatlimab 160mg — Neoadjuvant for 2 doses on days 1 and 29
  Other Names: Arm C
  Arms: Treatment Arm C
Drug: Ipilimumab 1mg/kg and nivolumab 3mg/kg — Neoadjuvant for 2 doses at days 1 and 22
  Other Names: Arm D (Cohort 1a)
  Arms: Treatment Arm D (Cohort 1a); Treatment Arm E (Cohort 1b)
Drug: Pembrolizumab 200 mg — Neoadjuvant for 2 doses at days 1 and 22
  Other Names: Arm F
  Arms: Treatment Arm F

SUMMARY:
This clinical trial is for patients with stage 3 cutaneous melanoma and patients with mucosal melanoma who are able to have surgery to remove all tumour deposits. To improve the chance that melanoma will not recurr, new experimental combinations of a type of treatment called immunotherapy will be given before surgery.

DETAILED DESCRIPTION:
This clinical trial is for patients with cutaneous melanoma which has spread to the lymph nodes (known as stage 3 melanoma) and for patients with any stage of mucosal melanoma. The study is for those patients who have disease that can be surgically removed.

The standard treatment for these patients is surgery to remove the affected tumour, lymph nodes, and any other deposits of melanoma, followed by drug therapy (known as adjuvant therapy). The most common drug therapy used to treat melanoma after surgery is known as 'immunotherapy'. Immunotherapy works by boosting the body's own immune system to better recognise and kill cancer cells.

The aim of the study is to offer new immunotherapy combinations to 3 cohorts of patients who are known to be poor responders to standard immunotherapy regimens.

Three cohorts of patients will be included:

1. Patients with resectable stage 3 cutaneous melanoma who have a predictive biomarker test result that indicates:

   Cohort 1a - they will be poor responders to standard anti-PD-1 immunotherapy (n=168) Cohort 1b - they will be high responders to standard anti-PD-1 immunotherapy (n=~154)
2. Patients with resectable stage 3 cutaneous melanoma who have had a recurrence of melanoma despite having standard anti-PD-1 based immunotherapy (n=111).
3. Patients with resectable mucosal melanoma, at any stage of disease. Mucosal melanoma is known to respond poorly to stabdard immunotherapy (n=60).

This research will test 6 combinations of immunotherapy which are given before surgery. Treatment given before surgery is known as 'neoadjuvant' treatment. Neoadjuvant treatment is standard for many cancers, including melanoma. The purpose of neoadjuvant immunotherapy is to increase the body's natural immune response by training it to recognise the evasive cancer cells before they are removed at surgery, and to shrink or destroy the melanoma, which may make surgery easier. This has been shown to reduce the chance of melanoma recurring after surgery. The drugs used in this study are called 'nivolumab', 'relatlimab', and 'ipilimumab' and 'pembrolizumab'

In this trial, there are 5 different study treatment combinations. Each combination uses different mechanisms to potentially overcome the predicted resistance to standard immunotherapy. There are 4 phases to the study:

1. Neoadjuvant treatment with one of the new immunotherapy combinations
2. Surgery
3. Adjuvant treatment with standard immunotherapy, IF the neoadjuvant therapy has not been effective enough to clear more than 10% of cancer cells.
4. Follow up for recurrence and survival to the end of 10 years

The main goal is to learn which of the new immunotherapy combinations are most effective at destroying the melanoma cells before surgery for each cohort of patients.

The other important goals are to learn which treatment is best at preventing the return of melanoma over 10 years and which increases survival from melanoma. The investigators also want to evaluate the side effects patients may have to treatment and how this affects the quality of life. The investigators will also continue to research biomarkers in blood, tumour tissue and stools to identify possible mechanisms for better response to therapy.

The study will be conducted in Australia and a total of 493 patients will be involved.

ELIGIBILITY:
COMMON Inclusion Criteria Applicable to all 3 cohorts

Inclusion Criteria:

* 1. Written informed consent
* 2. Male or female patients who are at least 18 years of age on the day of signing informed consent.
* 3. Clinically detectable disease, and/or RECIST version 1.1 defined disease, and/or disease confirmed on PET imaging.
* 4. Fully resectable disease defined as having no significant vascular, central nervous system or bony involvement. Only cases where a complete surgical resection leading to tumour free margins and which is safely achieved is considered "resectable".
* 5. Concurrent primary disease and lymph node metastases acceptable provided completely resectable.
* 6. Up to 3 in-transit metastases are permitted as long as these are fully resectable.
* 7. Tumour that is amenable to a newly obtained core biopsy for performance of the multi-omic predictive biomarker model
* 8. ECOG performance status of 0 to 1.
* 9. Adequate haematological, hepatic, renal and endocrine function
* 10. An anticipated life expectancy of >12 months.
* 11. Women of child bearing potential (WOCBP) must agree to avoid pregnancy or breast feeding for the duration of study treatment.

Inclusion Criteria - Cohort 1 only

* a. Histologically confirmed diagnosis of cutaneous melanoma or unknown primary melanoma
* b. AJCC 8th Ed Stage IIIB, IIIC, IIID cutaneous melanoma
* c. No prior systemic treatment for cutaneous melanoma
* d. Completion of the multi-omic predictive biomarker model within 14 days (7-10 business days) of planned randomisation.

Inclusion Criteria - Cohort 2 only

* a. Histologically confirmed diagnosis of cutaneous melanoma or unknown primary melanoma
* b. AJCC 8th Ed Stage IIIB, IIIC, IIID cutaneous melanoma
* c. Disease progression on neoadjuvant anti-PD-1 monotherapy, where progressed disease is completely resectable or, disease recurrence on adjuvant anti-PD-1 monotherapy, where recurrent disease is completely resectable
* d. No prior treatment with CTLA-4 or LAG-3 inhibitors.

Inclusion Criteria - Cohort 3 only

* a. Histologically confirmed diagnosis of mucosal melanoma
* b. Any stage of disease provided it is fully resectable
* c. No prior systemic treatment for mucosal melanoma

COMMON Exclusion Criteria Applicable to all 3 cohorts

* 1. Uveal melanoma
* 2. Any contraindication to the administration of relatlimab, ipilimumab or nivolumab
* 3. No prior systemic therapy, including treatment with prior anti-PD1/L1, anti-CTLA-4 or anti-LAG-3 therapy (cohorts 1 and 3), except for cohort 2 which will have received anti-PD1 monotherapy only.
* 4. A diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 14 days of randomisation. The following are permitted:

  1. Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc)
  2. Inhaled or intranasal corticosteroids (with minimal systemic absorption) may be continued if patient is on a stable dose
  3. Non-absorbed intra-articular steroid injections.
* 5. An active autoimmune disease that has required systemic treatment in the past 12 months (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). The following are permitted:

  1. Vitiligo
  2. Type I diabetes mellitus
  3. Residual autoimmune hypothyroidism on stable hormone replacement
  4. Resolved childhood asthma or atopy
  5. Psoriasis not requiring systemic treatment
  6. Autoimmune conditions which are not expected to recur in the absence of an external trigger.
* 6. A known additional malignancy that is progressing or has required active treatment within the past 3 years. The following malignancies, if undergone successful definitive resection or curative treatment, are permitted:

  1. Basal cell carcinoma of the skin
  2. Squamous cell carcinoma of the skin
  3. Carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy)
  4. Prostatic intraepithelial neoplasia
  5. In situ melanoma
  6. Atypical melanocytic hyperplasia
  7. Multiple primary melanomas
  8. Other malignancies for which the patient has been disease free for 1 year.
* 7. A known CNS metastases and/or carcinomatous meningitis
* 8. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis or current interstitial lung disease.
* 9. Has an active infection requiring systemic therapy.
* 10. Has a known history of Human Immunodeficiency Virus (HIV). Note: no testing for HIV is required unless mandated by local health authority.
* 11. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
* 12. Has a known history of active TB (Bacillus Tuberculosis).
* 13. Uncontrolled or significant cardiovascular disease including, but not limited to any of the following:

  1. Myocardial infarction (MI) or stroke/transient ischemic attack within the 6 months prior to consent
  2. Uncontrolled angina within the 3 months prior to consent
  3. Any history of clinically significant arrhythmias (such as poorly controlled atrial fibrillation, ventricular tachycardia, ventricular fibrillation, or torsades de pointes)
  4. QTc prolongation > 480 ms
  5. History of other clinically significant cardiovascular disease (i.e. cardiomyopathy, congestive heart failure with New York Heart Association functional classification III-IV, pericarditis, significant pericardial effusion, significant coronary stent occlusion, poorly controlled venous thrombosis, etc)
  6. Cardiovascular disease-related requirement for daily supplemental oxygen
  7. History of 2 or more M.I.s OR 2 or more coronary revascularisation procedures (regardless of the number of stent placements during each procedure)
  8. Patients with history of myocarditis, regardless of aetiology.
* 14. Patients with a >1+ proteinuria on urine dipstick testing unless a 24-hour urine collection for quantitative assessment indicates that the urine protein is <1 g/24 hours.
* 15. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the treating investigator.
* 16. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* 17. Pregnant or breast feeding females
* 18. Concurrent medical or social conditions that may prevent the patient from attending assessments per schedule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 494 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2038-01 (Estimated)

PRIMARY OUTCOMES:
Pathological response rate | Week 6
  The primary endpoint is the pathological response rate at surgery (between days 43 and 56) from the first dose of neoadjuvant study treatment for each of cohorts 1b, 2 and 3. The pathological response is categorised thus: - Complete pathological response (pCR) - 0% viable tumour cells in the surgical specimen - Near complete pathological response - (near pCR) - <10% viable tumour - Partial pathological response (pPR) - 10%-50% viable tumour - No pathological response (pNR) - >50% viable tumour The proportion of participants with a pCR, or near pCR will determine the pathological response rate.

SECONDARY OUTCOMES:
Event-free survival (EFS) | 10 years
  The proportion of patients with the earliest EFS outcome of: (a) Melanoma progression from randomisation and prior to planned surgery (b) Disease recurrence, from the date of surgery (local, regional or distant). (c) Study treatment-related death from randomisation. (d) Melanoma-related death, from randomisation.
Objective response rate | Week 6
  RECIST version 1.1 defined objective response at week 6 for patients with RECIST-measurable disease at baseline
Metabolic response rate | Week 6
  PERCIST defined metabolic response
Loco-regional relapse-free survival | 10 years
  Time from surgery to the date of loco-regional recurrence
Distant metastases-free survival | 10 years
  Time from surgery to the earliest date of distant recurrence, treatment-related death, or melanoma-related death
Overall survival | at 1, 2, 5 and 10 years
  Time from randomisation to death
Type, frequency and severity of drug-related toxicities | 30 days from last dose of study treatment
  The number, type, and grade of treatment-related adverse events per CTCAE version 5.0
Surgical adverse outcomes | At 3, 12 and 48 weeks post-operatively
  The number and grade of surgical complications according to the Clavien-Dindo Classification assessed at 3, 12 and 48 weeks post-operatively
Health related quality of life | 1 year
  The individual, summary and composite scores obtained from the validated EUROQOL QLQ-C30, EQ-5D, FACT-M (questions M10 to M17)
Comparison of the actual pathologocal response to each immunotherapy arm with the predicted pathological response to neoadjuvant immunotherapy based on the multi-omic predictive biomarker model | Week 6
  Correlation of the actual pathological response with the predicted response to combination neoadjuvant immunotherapy based on the multi-omic predictive biomarker model

CONTACTS AND LOCATIONS:
Overall Officials: Georgina Long, Study Chair — Melanoma Institute Australia
Locations (1):
- Melanoma Institute Australia, Wollstonecraft, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Undecided